CLINICAL TRIAL: NCT03482232
Title: Consequences of Doing What Should Not be Done in Primary Care
Acronym: SOBRINA
Status: Completed | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Osasunbidea (Unknown); Servicio Madrileño de Salud, Madrid, Spain (Other); Fondo de Investigacion Sanitaria (Other); AQuAS (Unknown); Agencia de Calidad Sanitaria de Andalucía (Unknown); Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government); Servicio Aragones De Salud (Other); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other); Generalitat Valenciana (Other); MurciaSalud (Other Government); Osakidetza (Other); Castilla-La Mancha Health Service (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: PI16/00816
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Overdose; Adverse Event
Keywords: patient safety; quality assurance; overuse
MeSH Terms: conditions — Drug Overdose | interventions — Benzodiazepines; Acetaminophen; Anti-Infective Agents; Anti-Bacterial Agents; Hypolipidemic Agents; Expectorants; Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients visiting GP: All patients visiting GP. The frequency of some drugs and diagnosis tests include in the Do-Not-Do recommendations will be analyzed.
  Interventions: Drug: Benzodiazepines; Drug: Non-steroidal anti-inflammatory drugs; Drug: paracetamol; Drug: Antimicrobial agent; Drug: Lipid-lowering drug; Diagnostic Test: Prostate cancer; Radiation: Lumbago
- Patient visiting pediatricians: All patients visiting pediatricians (0 to 14 years old). The frequency of some drugs and diagnosis tests include in the Do-Not-Do recommendations will be analyzed.
  Interventions: Drug: Antimicrobial agent; Drug: Mucolytic; Drug: Ibuprofen and paracetamol

INTERVENTIONS:
Drug: Benzodiazepines — Benzodiazepines for insomnia, agitation or delirium in people older than 65
  Groups: Patients visiting GP
Drug: Non-steroidal anti-inflammatory drugs — Non-steroidal anti-inflammatory drugs in patients with cardiovascular disease, chronic kidney disease, hypertension, heart failure or liver cirrhosis
  Groups: Patients visiting GP
Drug: paracetamol — paracetamol 1g for more than 3 days
  Groups: Patients visiting GP
Drug: Antimicrobial agent — antibiotic in acute bronchitis when the patient does not suffer from COPD, heart failure, diabetes or kidney disease or is undergoing active chemotherapy
  Other Names: Antibiotics
  Groups: Patients visiting GP
Drug: Lipid-lowering drug — Lipid-lowering drugs in patients older than 75 years without previous cardiovascular events
  Groups: Patients visiting GP
Diagnostic Test: Prostate cancer — Screening for prostate cancer in asymptomatic patients
  Groups: Patients visiting GP
Radiation: Lumbago — image tests in non-specific lumbago
  Groups: Patients visiting GP
Drug: Antimicrobial agent — antibiotics for pharyngitis (infants)
  Other Names: Antibiotics
  Groups: Patient visiting pediatricians
Drug: Mucolytic — mucolytics, antitussives or antibiotics for upper respiratory infections (infants)
  Other Names: Mucolytics
  Groups: Patient visiting pediatricians
Drug: Ibuprofen and paracetamol — treatment with ibuprofen and paracetamol (infants)
  Groups: Patient visiting pediatricians

SUMMARY:
Retrospective observational study in a random selection of 5% of digital records active between 2014 and 2017 to quantify the frequency of Do not do primary care recommendations, calculating the over-cost related to them and study reviewing a random selection of cases previously identified to determine whether patient suffered adverse events and their over-cost.

DETAILED DESCRIPTION:
Basement: Overuse subjected patients to unnecessary risk without promoting a sufficient clinical benefit and over-cost. The Less is More Medicine movement has led to the identification of Do not do in different specialties, also in primary care.

Objective: To analyze the impact of errors (overuse rates based in Do not do recommendations) in clinical practice.

Method: Retrospective observational study in a random selection of 5% of digital records active between 2014 and 2017 to quantify the frequency of Do not do primary care recommendations, calculating the over-cost related to them. Retrospective study reviewing a random selection of cases previously identified to determine whether patient suffered adverse events and their over-cost.

Setting. Primary care in Andalucía, Aragón, Castilla La Mancha, Comunidad Valenciana, Madrid, Murcia, Navarra y País Vasco, eight autonomous communities in Spain.

ELIGIBILITY:
Inclusion Criteria:

* All patients visiting GPs

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients data codified in the primary care databases (BDCAP and BIFAP)
Sampling Method: Non-Probability Sample
Enrollment: 750000 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Medical overuse | Three years
  Inadequate prescriptions of antimicrobials, mucolytics, lipid-lowering-drugs, ibuprofen or paracetamol in some specific cases defined as overuse
Medical overuse | Three years
  Inadequate test for lumbalgia or prostate cancer

SECONDARY OUTCOMES:
Adverse events as consequence of inadequate clinical decision [Safety] | Three years
  Patients suffering hurt due to inadequate prescription or inadequate test. Inadequate prescriptions or tests as defined by Do-not-Do recommendations. These were defined by Spanish Primary Care Scientific Societies

CONTACTS AND LOCATIONS:
Overall Officials: JOSE J MIRA, PhD, Principal Investigator — UNIVERSIDAD MIGUEL HERNANDEZ
Locations (2):
- Spain (2):
  - FISABIO, Elche, Alicante
  - Universidad Miguel Hernández, Elche, Alicante

IPD SHARING:
Plan to Share IPD: Yes
Public and safety patient researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2019
Access Criteria: http://www.nohacer.es
URL: http://www.nohacer.es

REFERENCES:
- [Background] Gibson R. The human cost of overuse. BMJ. 2014 May 6;348:g2975. doi: 10.1136/bmj.g2975. No abstract available. PMID 24803401
- [Background] Brownlee S, Chalkidou K, Doust J, Elshaug AG, Glasziou P, Heath I, Nagpal S, Saini V, Srivastava D, Chalmers K, Korenstein D. Evidence for overuse of medical services around the world. Lancet. 2017 Jul 8;390(10090):156-168. doi: 10.1016/S0140-6736(16)32585-5. Epub 2017 Jan 9. PMID 28077234
- [Background] Segal JB, Bridges JF, Chang HY, Chang E, Nassery N, Weiner J, Chan KS. Identifying possible indicators of systematic overuse of health care procedures with claims data. Med Care. 2014 Feb;52(2):157-63. doi: 10.1097/MLR.0000000000000052. PMID 24374418
- [Background] Rosenberg A, Agiro A, Gottlieb M, Barron J, Brady P, Liu Y, Li C, DeVries A. Early Trends Among Seven Recommendations From the Choosing Wisely Campaign. JAMA Intern Med. 2015 Dec;175(12):1913-20. doi: 10.1001/jamainternmed.2015.5441. PMID 26457643
- [Background] Grady D, Redberg RF. Less is more: how less health care can result in better health. Arch Intern Med. 2010 May 10;170(9):749-50. doi: 10.1001/archinternmed.2010.90. No abstract available. PMID 20458080
- [Background] Aranaz-Andres JM, Aibar C, Limon R, Mira JJ, Vitaller J, Agra Y, Terol E. A study of the prevalence of adverse events in primary healthcare in Spain. Eur J Public Health. 2012 Dec;22(6):921-5. doi: 10.1093/eurpub/ckr168. Epub 2011 Nov 29. PMID 23180803
- [Background] Newton EH, Zazzera EA, Van Moorsel G, Sirovich BE. Undermeasuring Overuse--An Examination of National Clinical Performance Measures. JAMA Intern Med. 2015 Oct;175(10):1709-11. doi: 10.1001/jamainternmed.2015.4025. No abstract available. PMID 26258406
- [Derived] Mira JJ, Carrillo I, Perez-Perez P, Astier-Pena MP, Caro-Mendivelso J, Olivera G, Silvestre C, Nuin MA, Aranaz-Andres JM; on behalf the SOBRINA Research Team. Avoidable Adverse Events Related to Ignoring the Do-Not-Do Recommendations: A Retrospective Cohort Study Conducted in the Spanish Primary Care Setting. J Patient Saf. 2021 Dec 1;17(8):e858-e865. doi: 10.1097/PTS.0000000000000830. PMID 34009877
- [Derived] Mira JJ, Carrillo I, Gea Velazquez de Castro MT, Silvestre C, Olivera G, Caro-Mendivelso J, Perez-Perez P, Agra Y, Fernandez AM, Aranaz-Andres JM; SOBRINA Research Team. SOBRINA Spanish study-analysing the frequency, cost and adverse events associated with overuse in primary care: protocol for a retrospective cohort study. BMJ Open. 2019 Mar 4;9(3):e023399. doi: 10.1136/bmjopen-2018-023399. PMID 30837247